CLINICAL TRIAL: NCT06169319
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled, Dose-ranging Study to Assess the Efficacy, Safety, and Tolerability of EN3835 vs Placebo in the Treatment of Plantar Fasciitis (PFA)
Brief Title: A Study to Assess Collagenase Clostridium Histolyticum (CCH) in the Treatment of Plantar Fasciitis (PFA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3835-227
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Microbial Collagenase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: CCH High Dose (Experimental): Participants will receive a high dose of CCH on Day 1.
  Interventions: Biological: Collagenase Clostridium Histolyticum (CCH)
- Group 2: CCH Low Dose (Experimental): Participants will receive a low dose of CCH on Day 1.
  Interventions: Biological: Collagenase Clostridium Histolyticum (CCH)
- Group 3: Placebo (Placebo Comparator): Participants will receive matching placebo on Day 1.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Collagenase Clostridium Histolyticum (CCH) — Biologic: Intrafascial injection
  Other Names: EN3835
  Arms: Group 1: CCH High Dose; Group 2: CCH Low Dose
Biological: Placebo — Intrafascial injection
  Arms: Group 3: Placebo

SUMMARY:
This study will assess the efficacy, safety, and tolerability of 2 different doses of collagenase clostridium histolyticum (CCH) (previously known as EN3835) compared to placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Have no significant medical history or examination findings related to the foot to be treated, which in the investigator's opinion, would make the participant unsuitable for study intervention administration.
* Have a diagnosis of plantar fasciitis for ≥6 months, which has not responded to conservative therapies. Conservative therapies may include rest, physical therapy, splinting/bracing, orthotics, icing, physiotherapy, acetaminophen, corticosteroids, or nonsteroidal anti-inflammatory drugs (NSAIDs).
* Have current foot pain due to plantar fasciitis.

Key Exclusion Criteria:

* Has any musculoskeletal, neuromuscular, neurosensory, other neurological or related disorder that affects the participant's use of his/her feet and/or would impair his/her completion of study assessments as determined by the investigator either due to the disorder or due to pain.
* Has a clinically meaningful laboratory abnormality.
* Has a body mass index ≥35 kilograms per meter squared (kg/m^2).
* Has a known bleeding disorder, which, in the investigator's opinion, would make the participant unsuitable for enrollment in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline at Week 12 in the Weekly Mean of the Average Daily (24-hour) Pain (ADP) Score as Measured on the Pain Intensity Numeric Rating Scale (NRS) | Baseline, Week 12

SECONDARY OUTCOMES:
Change from Baseline up to Day 85 in the Foot Function Index (FFI) Difficulty Subscale Score | Baseline, up to Day 85
Change from Baseline up to Day 85 in the FFI Activity Limitation Subscale Score | Baseline, up to Day 85
Change from Baseline up to Week 12 in the Weekly Mean of the ADP Score as Measured on the Pain Intensity NRS | Baseline, up to Week 12
Change from Baseline up to Day 85 in the FFI Pain Subscale Score | Baseline, up to Day 85
Change from Baseline up to Day 85 in the FFI Total Score | Baseline, up to Day 85
Number of Participants That Used Rescue Analgesic Medication | Up to Day 85
Total Amount (milligrams [mg]) of Rescue Analgesic Medication Used | Up to Day 85
Patient Global Impression of Change (PGIC) Foot Pain Scale Score | Up to Day 85
Clinician Global Impression of Change (CGIC) Scale Score | Up to Day 85
Subject Satisfaction with Treatment Scale Score | Up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Endo Pharmaceuticals
Locations (39):
- United States (39):
  - Endo Site 8, Tucson, Arizona
  - Endo Site 20, Castro Valley, California
  - Endo Site 13, Corona, California
  - Endo Site 6, Encinitas, California
  - Endo Site 11, Fresno, California
  - Endo Site 16, Los Angeles, California
  - Endo Site 40, Los Angeles, California
  - Endo Site 21, San Francisco, California
  - Endo Site 10, Tarzana, California
  - Endo Site 37, Coconut Creek, Florida
  - Endo Clinical Site 3, Pinellas Park, Florida
  - Endo Site 14, Sweetwater, Florida
  - Endo Site 7, Lawrenceville, Georgia
  - Endo Site 23, Stonecrest, Georgia
  - Endo Site 31, North Chicago, Illinois
  - Endo Site 28, O'Fallon, Illinois
  - Endo Site 33, Overland Park, Kansas
  - Endo Site 35, Shreveport, Louisiana
  - Endo Clinical Site 2, Pasadena, Maryland
  - Endo Site 19, Grand Rapids, Michigan
  - Endo Site 27, Missoula, Montana
  - Endo Site 38, Westwood, New Jersey
  - Endo Site 25, Moore, Oklahoma
  - Endo Site 39, Portland, Oregon
  - Endo Site 36, Malvern, Pennsylvania
  - Endo Clinical Site 4, Bedford, Texas
  - Endo Site 24, Burleson, Texas
  - Endo Site 17, Dallas, Texas
  - Endo Site 26, Dallas, Texas
  - Endo Site 18, Dallas, Texas
  - Endo Site 30, Fort Worth, Texas
  - Endo Clinical Site 1, Georgetown, Texas
  - Endo Site 15, Houston, Texas
  - Endo Site 9, McAllen, Texas
  - Endo Site 34, San Antonio, Texas
  - Endo Site 22, San Antonio, Texas
  - Endo Clinical Site 5, Salt Lake City, Utah
  - Endo Site 32, Newport News, Virginia
  - Endo Site 12, Suffolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP